CLINICAL TRIAL: NCT03936764
Title: Effect of Two Different Preoperative Training Densities in Patients With Non-small-cell Lung Cancer Before Lung Resection Surgery
Acronym: Preo-Dens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Preo-Dens; ID-RCB : 2018-A03301-54 (Registry Identifier: 2018-A03301-54)
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Preoperative pulmonary rehabilitation; Preoperative training; Prehabilitation; Lung resection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): 5 Preoperative Pulmonary Rehabilitation sessions / week during 3 weeks.
  Interventions: Other: Preoperative Pulmonary Rehabilitation
- Group 2 (Other): 3 Preoperative Pulmonary Rehabilitation sessions / week during 5 weeks.
  Interventions: Other: Preoperative Pulmonary Rehabilitation

INTERVENTIONS:
Other: Preoperative Pulmonary Rehabilitation — Each prehabilitation session will last approximately 90 minutes and will include:
  * Endurance training at the ventilatory threshold, determined according to the initial CPET. The first session will last for 15 to 20 minutes then increase by 5 minutes each session to reach 45 minutes in total (including a 5-minute warm-up and 5 minutes of active recovery). The intensity will then increase by 5 or 10 W, as could be tolerated;
  * Peripheral muscle strengthening at 60% to 70% of the 1-repetition maximum of 3 main components (quadriceps press, whole-leg extension, and upper limb pull down). Three sets of 12 movements will carry out for each exercise and the load will increase weekly as tolerated;
  * Inspiratory muscle training using a threshold calibrated to at least 30% of the MIP. Patients will be encouraged to carry out 15 minutes of independent training daily and to increase the resistance regularly.
  * Education to bronchial drainage techniques as well as directed coughing.

SUMMARY:
Pulmonary resection surgery is currently the recommended curative treatment for early stages of non-small cell lung cancer. The implementation of preoperative respiratory rehabilitation programs has shown beneficial results on pulmonary function, functional level, cardiorespiratory conditioning and the occurrence and severity of postoperative complications in this population of patients. Despite these benefits, the most recent meta-analyzes highlight the fact that training modalities (duration, frequencies, intensity) are very heterogeneous. It is then difficult to structure a program only on the basis of data from the literature.

In a cohort analysis of 50 patients trained from 2014 to 2017, our team reported a significantly greater improvement in physiological parameters in patients who performed 15 or more preoperative training sessions. This number of 15 outpatient sessions is therefore considered a minimum training goal in our current practice.

The difficulty of the oncological context is to find the compromise between the necessary diligence to initiate the cancer surgical treatment and the necessary time to obtain the benefits of the preoperative rehabilitation. Previous study reports the difficulty of setting up a four-week training program, perceived as delaying surgery. In order to prevent any risk of prolonging the surgical management time, rehabilitation teams routinely offer short programs with high training frequencies of up to five to six sessions per week. It seems important to note that preoperative rehabilitation is normally considered in patients for whom there is a risk of moderate to high postoperative complications according to the European and North American recommendations. Thus these patients generally benefit from a longer period of assessment than patients whose risk is considered low in terms of their cardio-respiratory and muscular function.

The median duration between the physiological evaluation of patients considered "at risk" before pulmonary resection surgery is 44 (Q1-Q3 29-76) days at Rouen University Hospital, with no significant differences observed between patients who have benefited or not from preoperative rehabilitation. Some teams have even pointed out that there is no difference in survival prognosis in the short or long term between patients who have had an operative delay of more or less 60 or 90 days respectively, which shows the compatibility with the set up a dedicated training course.

As mentioned earlier, the concept of delay has led to extremely dense training for a functionally and cardio-respiratory fragile target population as evidenced by pejorative VO2peak. The density of the training, failing to generate significant physiological stimulation, may increase fatigue or limit adherence to training, especially if it requires movement, and is added to a therapeutic planning including many consultations and further examinations. To date, no study has evaluated the density of preoperative supervised training on pre-surgical benefits.

The objective of this work is to compare the effectiveness of a program of 15 training sessions on VO2peak according to two different densities, namely five times a week over three weeks, or three times a week over five weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old;
* Beneficiary of a social security scheme;
* Non-Small Cell Lung Cancer or suspicion of bronchial neoplasia;
* Addressed to respiratory rehabilitation in a preoperative setting with a moderate to high risk estimate (VO2peak < 20 ml/kg/min);
* Intervention date not established when included in the program or ≥ 5 wk.

Exclusion Criteria:

* Patient under guardianship;
* Pregnant or lactating woman;
* Cardiological contraindication to training;
* Neoadjuvant radio-chemotherapy;
* Refusal to carry out a training program in a rehabilitation center;
* Orthopedic, neurological, vascular or neuromuscular pathology limiting training;
* Exacerbation or deterioration of the general condition requiring stopping the preoperative re-training program;
* Modification of the therapeutic project at a multidisciplinary consultation meeting requiring the cessation of rehabilitation or participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
peak dioxyen consumption (VO2peak) | before the preoperative training program
  VO2peak (in ml/kg/min) measured during and incremental Cardio-Pulmonary Exercise Testing (CPET)
peak dioxyen consumption (VO2peak) | through preoperative training program completion (15 sessions)
  VO2peak (in ml/kg/min) measured during and incremental Cardio-Pulmonary Exercise Testing (CPET)

SECONDARY OUTCOMES:
peak work-rate (WRpeak) | before the preoperative training program
  maximum power reached during the Cardio-Pulmonary Exercise Testing (CPET)
peak work-rate (WRpeak) | through preoperative training program completion (15 sessions)
  maximum power reached during the Cardio-Pulmonary Exercise Testing (CPET)
oxygen consumption at ventilatory threshold (VO2vt) | before the preoperative training program
  oxygen consumption at ventilatory threshold recorded during the Cardio-Pulmonary Exercise Testing (CPET)
oxygen consumption at ventilatory threshold (VO2vt) | through preoperative training program completion (15 sessions)
  oxygen consumption at ventilatory threshold recorded during the Cardio-Pulmonary Exercise Testing (CPET)
work-rate at ventilatory threshold (WRvt) | before the preoperative training program
  work-rate at ventilatory threshold recorded during the Cardio-Pulmonary Exercise Testing (CPET)
work-rate at ventilatory threshold (WRvt) | through preoperative training program completion (15 sessions)
  work-rate at ventilatory threshold recorded during the Cardio-Pulmonary Exercise Testing (CPET)
ventilatory efficiency (VE/VCO2 slope) | before the preoperative training program
  linear regression of the ratio between the increase in minute ventilation and the expired carbon dioxide flow (VE/VCO2 slope)
ventilatory efficiency (VE/VCO2 slope) | through preoperative training program completion (15 sessions)
  linear regression of the ratio between the increase in minute ventilation and the expired carbon dioxide flow (VE/VCO2 slope)
body mass index (BMI) | before the preoperative training program
  weight in kilograms divided by the square of height in meters
body mass index (BMI) | through preoperative training program completion (15 sessions)
  weight in kilograms divided by the square of height in meters
fat-free mass | before the preoperative training program
  impedancemetry (Bodystat® 1500MDD, (5/50 kHz), Bodystat, Douglas, Isle of Man, UK).
fat-free mass | through preoperative training program completion (15 sessions)
  impedancemetry (Bodystat® 1500MDD, (5/50 kHz), Bodystat, Douglas, Isle of Man, UK).
quadriceps peak torque | before the preoperative training program
  quadriceps peak torque (in Nm) assessed by dynamometry (MicroFET2®, Hogan Health Industries, Inc., UT)
quadriceps peak torque | through preoperative training program completion (15 sessions)
  quadriceps peak torque (in Nm) assessed by dynamometry (MicroFET2®, Hogan Health Industries, Inc., UT)
maximum inspiratory pressure (MIP) | before the preoperative training program
  Maximum negative oral pressure generated by the patient during inspiration (in cmH2O)
maximum inspiratory pressure (MIP) | through preoperative training program completion (15 sessions)
  Maximum negative oral pressure generated by the patient during inspiration (in cmH2O)
Health related quality of life (HRQoL) questionnaire | before the preoperative training program
  Full name of the scale : "European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire and modular supplement for Lung Cancer patients" (EORTC QLQ-C30 / LC13) The EORTC QLQ-C30, is a 30 questions questionnaire developed by the European Organization for Research and Treatment of Cancer, to assess the QoL of cancer patients. It has been translated and validated into over 100 languages and is used in more than 3,000 studies worldwide.
  For patients with Lung Cancer, a 13 questions modular supplement, the LC-13, is validated.
  The HRQoL is therefore evaluated by a set of 43 questions gathering all aspects that could be impacted.
  A raw score is calculated for each dimension and summary score, then standardized from 0 to 100 points. The additional module for Lung Cancer (LC-13) provides a complementary dimension with specific items related to the tumor site.
  (see Fayers et. al., The EORTC QLQ-C30 Scoring Manual (3rd Edition) 2001.
Health related quality of life (HRQoL) questionnaire | through preoperative training program completion (15 sessions)
  Full name of the scale : "European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire and modular supplement for Lung Cancer patients" (EORTC QLQ-C30 / LC13) The EORTC QLQ-C30, is a 30 questions questionnaire developed by the European Organization for Research and Treatment of Cancer, to assess the QoL of cancer patients. It has been translated and validated into over 100 languages and is used in more than 3,000 studies worldwide.
  For patients with Lung Cancer, a 13 questions modular supplement, the LC-13, is validated.
  The HRQoL is therefore evaluated by a set of 43 questions gathering all aspects that could be impacted.
  A raw score is calculated for each dimension and summary score, then standardized from 0 to 100 points. The additional module for Lung Cancer (LC-13) provides a complementary dimension with specific items related to the tumor site.
  (see Fayers et. al., The EORTC QLQ-C30 Scoring Manual (3rd Edition) 2001.
Adherence to sessions | through preoperative training program completion (15 sessions)
  number of sessions performed on number of sessions planned
Postoperative Complications | At 30 days post-intervention
  number and type of complication during the 30 days post lung resection. Each complication severity is evaluated with the Clavien-Dindo scale.

CONTACTS AND LOCATIONS:
Locations (1):
- ADIR Association, Bois-Guillaume, Normandy, France

REFERENCES:
- [Derived] Gravier FE, Smondack P, Boujibar F, Prieur G, Medrinal C, Combret Y, Muir JF, Baste JM, Cuvelier A, Debeaumont D, Bonnevie T. Prehabilitation sessions can be provided more frequently in a shortened regimen with similar or better efficacy in people with non-small cell lung cancer: a randomised trial. J Physiother. 2022 Jan;68(1):43-50. doi: 10.1016/j.jphys.2021.12.010. Epub 2021 Dec 21. PMID 34952813